CLINICAL TRIAL: NCT02772419
Title: A Phase 2, Double-Blind, Placebo-Controlled Study of Benralizumab (KHK4563) in Patients With Eosinophilic Chronic Rhinosinusitis
Brief Title: Study of Benralizumab (KHK4563) in Patients With Eosinophilic Chronic Rhinosinusitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4563-005
Record Dates: First submitted 2016-04-25; First posted 2016-05-13 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Eosinophilic Chronic Rhinosinusitis
MeSH Terms: interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- benralizumab A (Experimental): Subcutaneous (SC) administration
  Interventions: Drug: benralizumab
- benralizumab B (Experimental): SC administration
  Interventions: Drug: benralizumab
- Placebo (Placebo Comparator): Placebo SC administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: benralizumab — SC administration
  Arms: benralizumab A
Drug: benralizumab — SC administration
  Arms: benralizumab B
Drug: Placebo — SC administration
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of SC administrations of Benralizumab or Placebo in the subjects with Eosinophilic Chronic Rhinosinusitis in a multicenter, randomized, double-blind, placebo-controlled study. The pharmacokinetics and immunogenicity will be assessed secondarily.

DETAILED DESCRIPTION:
Screening Period (maximum 4 weeks) , Randomized Treatment Period (24 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Patients 20 years to 75 years of age
* Eosinophilic chronic rhinosinusitis with a total score of ≥ 11 according to the diagnosis of eosinophilic chronic rhinosinusitis at enrollment
* A minimum bilateral nasal polyp score of 3 out of the maximum score of 8 (with a score of at least 1 out of the maximum score of 4 for each nostril) at screening and at enrollment
* Weight of ≥ 40 kg at screening

Exclusion Criteria:

* A Sino-Nasal Outcome Test-22 (SNOT-22) score of < 7 at enrollment
* Any nasal surgery (including polypectomy) within 1 year prior to the date of consent
* Hospitalization for ≥ 24 hours for treatment of asthma exacerbation, within 12 weeks prior to the date of consent
* Exposure to any commercially available (e.g., omalizumab) or investigational biologic agent within 16 weeks or 5 half-lives prior to enrollment, whichever is longer
* Use of systemic corticosteroids (including oral corticosteroids) or corticosteroid nasal solution (except spraying) within 4 weeks prior to enrollment or planned use of such medications during the double-blind period
* Prior treatment with benralizumab

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
The change from baseline in nasal polyp score at Week 12 | baseline and 12 weeks post-dose

SECONDARY OUTCOMES:
The change from baseline in nasal polyp score | Pre-dose and 4,8,12,16,20,24 weeks post-dose
The change from baseline in Computed tomography (CT) score | baseline and 12 weeks post-dose
Number of subjects discontinued from the study due to aggravation of eosinophilic chronic rhinosinusitis | Up to 24 weeks after dosing
Time to discontinuation (days) from the study due to aggravation of eosinophilic chronic rhinosinusitis | Up to 24 weeks after dosing
The change from baseline in Blood eosinophil count | Pre-dose and 4,8,12,16,20,24 weeks post-dose
The change from baseline in Nasal Airway Resistance | Pre-dose and 4,8,12,24 weeks post-dose
  Nasal airway resistance (Pa/cm^3/s)
The change from baseline in the averaged values of the Olfactory thresholds | Pre-dose and 4,8,12,24 weeks post-dose
  Olfactory thresholds are assessed by T&T Olfactometer Test Score (Five kinds of smell with eight (5 to -2) phases).
The change from baseline in the improvement of olfactory dysfunction | Pre-dose and 4,8,12,24 weeks post-dose
  Olfactory dysfunction (1 to 5) is calculated by the Olfactory thresholds.
The change from baseline in Sino-Nasal Outcome Test-2 (SNOT-22) | Pre-dose and 4,8,12, 16, 20, 24 weeks post-dose
  Symptom score are assessed by VAS (nasal congestion, anterior and posterior nasal drip, loss of the sense of smell, headache, and impairment in activity of daily living)
The change from baseline in Symptom score by Visual Analog Scale (VAS) | Pre-dose and 4,8,12, 16, 20, 24 weeks post-dose
  Symptom score are assessed by VAS (nasal congestion, anterior and posterior nasal drip, loss of the sense of smell, headache, and impairment in activity of daily living)
Incidence of treatment-emergent adverse events (TEAEs) or drug-related TEAEs and their nature | Up to 24 weeks after dosing

OTHER OUTCOMES:
Serum concentration of benralizumab | Pre-dose and 4, 8, 12, 16, 20, 24 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tokunaga T, Sakashita M, Haruna T, Asaka D, Takeno S, Ikeda H, Nakayama T, Seki N, Ito S, Murata J, Sakuma Y, Yoshida N, Terada T, Morikura I, Sakaida H, Kondo K, Teraguchi K, Okano M, Otori N, Yoshikawa M, Hirakawa K, Haruna S, Himi T, Ikeda K, Ishitoya J, Iino Y, Kawata R, Kawauchi H, Kobayashi M, Yamasoba T, Miwa T, Urashima M, Tamari M, Noguchi E, Ninomiya T, Imoto Y, Morikawa T, Tomita K, Takabayashi T, Fujieda S. Novel scoring system and algorithm for classifying chronic rhinosinusitis: the JESREC Study. Allergy. 2015 Aug;70(8):995-1003. doi: 10.1111/all.12644. Epub 2015 May 26. PMID 25945591